CLINICAL TRIAL: NCT06947174
Title: The Role of Angiographic Measurements and Anatomical Correlations in Intra-Aortic Balloon Pump (IABP) Size Selection
Status: Recruiting | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, James Tisyakorn, Principle Investigator, Siriraj Hospital
Other Study IDs: 928/2567(IRB4)
Record Dates: First submitted 2025-04-07; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Intra-aortic Balloon Pump
Keywords: Intra-aortic balloon pump

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this study aim to accurately size the IABP size for patients. The main questions it aims to answer are:

* Are patients's height, jugular notch to transpyloric plane distance and distance from the carina to the upper part of the first lumbar vertebra (measured by chest X-ray) are a good surrogate for IABP sizing?
* Is the distance obtained during a transfemoral artery catheterization a reliable way to size the IABP? Researchers will enroll patient who have had previous CT that include thoracic aorta to celiac trunk who will undergo transfemoral angiography.
* All patients that researcher enrolled will undergo transfemoral angiography, during which the researchers will measure the vessel distance using a wire after the procedure end.
* Researchers will measure the height weight, jugular notch to transpyloric plane distance, CXR distance from carina to upper border of L1 and the distance from aorta at subclavian level to celiac trunk from CT.
* Researchers will find the correlation between of each measurement to the distance from aorta at subclavian level to celiac trunk from CT (considered the standard measure).

DETAILED DESCRIPTION:
Background:

* Intra-aortic balloon pumps (IABP) are commonly used as mechanical circulatory support in patient with cariogenic shock.
* Proper sizing of IABP is critical, critical, with the balloon typically extending from the left subclavian artery to the celiac axis, and occupying 90-95% of the aorta's diameter during each cycle.
* Manufacturers usually recommend balloon sizes based on patient height. However, previous studies suggest that the accuracy of these recommendations varies. One study found that while chest X-ray (CXR) confirmed correct balloon positioning in 96.8% of cases, only 38.1% were accurately positioned based on CT scans.
* Malposition of the balloon, such as blocking the renal or mesenteric arteries, may lead to complications like renal or intra-abdominal ischemia
* Cadaveric studies have suggested that the distance from the jugular notch to the transpyloric plane correlates more strongly with the subclavian-to-celiac artery distance than height alone
* A Chinese study attempted to predict the left subclavian artery to celiac trunk distance using a combination of height, body mass index (BMI), and age
* In this study, investigators want to find the better way in sizing IABP balloon. Investigators with use the height, age, weight, jugular notch to transpyloric plane distance, distance from the carina to the upper part of the first lumbar vertebra (measured by chest X-ray) and length of the vessel measured during transfemoral angiography compare with distance of the vessel measure during CT-scan.

Outcome

* Investigators will find the correlation between height, jugular notch to transpyloric plane distance, wire pull out distance from aortic knob to L1 in angiographic study and distance of left subclavian artery to celiac trunk measure from CT aorta using Pearson Correlation or Spearman rank statistics.
* Referencing previous studies

The correlation coefficient between height and the distance to the LCA-celiac trunk was 0.369 , and the correlation coefficient between height and the distance to the LCA-renal artery was 0.579 (Igari T. The length of the aorta from the subclavian artery to the renal artery based on computed tomographic measurements in Japanese adults. Journal of Artificial Organs. 2006;9:267-70.). The researcher chose to use the lower correlation coefficient of 0.369 for calculating sample size to achieve a maximum sample size.Using the formula for calculating sample size for correlation coefficient testing, with a standard value of 1.96 set at a significance level of 5% and a power of 80%, the sample size was calculated as follows:

* Fisher's Z Transformation from formula = = 1/2 ln((1+(0.369))/(1-(0.369)))= 0.387 Calculate sample size by n= ((1.96+0.84)/(0.387))^2+3 n = 56 Sample size from this calculation is 56, it was determined that an additional sample size of 56 participants is needed, with a further increase of 20% to account for potential data loss, resulting in an additional 12 participants, totaling 68 individuals. Therefore, the sample size used in this study is 68 participants Recruitments - Investigators will review patients scheduled for angiography to determine if they have had a CT chest scan that includes the celiac trunk and are eligible for the study.

Inclusion criteria are

1. Patient age ≥ 18 years old
2. Patients had obtained CT scan of chest with upper abdomen with celiac trunk visualize within 1 year from the day of transfemoral angiography
3. Patients had who will undergo transfemoral angiography as clinical indicated
4. Patients had obtained Chest X-ray within 1 year from the day of transfemoral angiography Exclusion criteria are

1. Patient with limb amputation 2. Patient with known aortic abnormalities such as aortic aneurysm, aortic dissection Study procedure

* Before the patient's arrival at the catheterization lab, the investigator will seek their consent to participate in the study.
* Patients will be informed that their treatment will proceed as usual, with the only additional step being a request for the procedure operator to measure the pullback wire distance at the end of the procedure. This step will result in slightly more radiation exposure but will take less than one minute to complete and does not increase the procedural risk.
* If the operator determines that the patient is unstable, the measurement will not be performed. Patients who choose not to participate will still receive their standard treatment without any changes.
* Other measurements such as height weight will be collected per Cath lab protocol.
* The measurement of jugular notch to transpyloric plane distance will be collect at the recovery ward.

ELIGIBILITY:
Inclusion Criteria:

* Patients had obtained CT scan of chest with upper abdomen with celiac trunk visualize within 1 year from the day of transfemoral angiography
* Patients had who will undergo transfemoral angiography as clinical indicated
* Patients had obtained Chest X-ray within 1 year from the day of transfemoral angiography

Exclusion Criteria:

* Patient with limb amputation
* Patient with known aortic abnormalities such as aortic aneurysm, aortic dissection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing transfemoral angiography at Siriraj cauterization lab.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Height | Day 1
  Height of the patients
Weight | Day 1
  Weight of the patient
Jugular notch to transpyloric plane distance | Day 1
  Distance from jugular notch to transpyloric plane (Horizontal plane between jugular notch to pubic symphysis)
distance from the carina to the upper part of the first lumbar vertebra (measured by chest X-ray) | through study completion, an average of 1 year
  distance from the carina to the upper part of the first lumbar vertebra (measured by chest X-ray)
distance of left subclavian artery to celiac trunk measure from CT scan. | through study completion, an average of 1 year
  distance of left subclavian artery to celiac trunk measure from CT scan.
distance from the carina to the upper part of the first lumbar vertebra measure by wiring distance during transferal angiography | Day 1
  Wiring distance is obtained during the transferal angiography after the procedure is done and when the operator take the wire out. Mesure at the carina level to the upper part of the first lumbar vertebra

CONTACTS AND LOCATIONS:
Overall Officials: Ploy Pengchata, Doctor of Medicine, Principal Investigator — Her Majesty Cardiac Center, Faculty of Medicine Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 years after the study end
Access Criteria: Data sharing upon reasonable request.

REFERENCES:
- [Background] Yang IY, Oraee S, Viejo C, Stern H. Computed tomography celiac trunk topography relating to celiac plexus block. Reg Anesth Pain Med. 2011 Jan-Feb;36(1):21-5. doi: 10.1097/AAP.0b013e318203067f. PMID 21455084
- [Background] Kim JT, Lee JR, Kim JK, Yoon SZ, Jeon Y, Bahk JH, Kim KB, Kim CS, Lim YJ, Kim HS, Kim SD. The carina as a useful radiographic landmark for positioning the intraaortic balloon pump. Anesth Analg. 2007 Sep;105(3):735-8. doi: 10.1213/01.ane.0000278086.23266.35. PMID 17717232
- [Background] Chaturvedi A, Rotman Y, Hoang T, Jew G, Mandalapu A, Narins C. CT and chest radiography in evaluation of mechanical circulatory support devices for acute heart failure. Insights Imaging. 2023 Jul 16;14(1):122. doi: 10.1186/s13244-023-01469-8. PMID 37454301
- [Background] Rhodes NG, Johnson TF, Boyum JH, Khandelwal A, Howell BD, Froemming AT, Behfar A. Radiology of Intra-Aortic Balloon Pump Catheters. Radiol Cardiothorac Imaging. 2022 Apr 14;4(2):e210120. doi: 10.1148/ryct.210120. eCollection 2022 Apr. PMID 35506140
- [Background] Parissis H, Soo A, Leotsinidis M, Dougenis D. A statistical model that predicts the length from the left subclavian artery to the celiac axis; towards accurate intra aortic balloon sizing. J Cardiothorac Surg. 2011 Aug 9;6:95. doi: 10.1186/1749-8090-6-95. PMID 21827666
- [Background] Byon HJ, Kim H, Kim HC, Kim JT, Kim HS, Lee SC, Kim CS. Potential risk for intra-aortic balloon-induced obstruction to the celiac axis or the renal artery in the Asian population. Thorac Cardiovasc Surg. 2011 Mar;59(2):99-102. doi: 10.1055/s-0030-1250429. Epub 2011 Mar 7. PMID 21384305
- [Background] Igari T. The length of the aorta from the subclavian artery to the renal artery based on computed tomographic measurements in Japanese adults. J Artif Organs. 2006;9(4):267-70. doi: 10.1007/s10047-006-0346-z. Epub 2006 Dec 21. PMID 17171407
- [Background] Shin H, Yozu R, Sumida T, Kawada S. Acute ischemic hepatic failure resulting from intraaortic balloon pump malposition. Eur J Cardiothorac Surg. 2000 Apr;17(4):492-4. doi: 10.1016/s1010-7940(00)00366-3. PMID 10773577
- [Background] Swartz MT, Sakamoto T, Arai H, Reedy JE, Salenas L, Yuda T, Standeven JW, Pennington DG. Effects of intraaortic balloon position on renal artery blood flow. Ann Thorac Surg. 1992 Apr;53(4):604-10. doi: 10.1016/0003-4975(92)90318-x. PMID 1554268
- [Background] Rastan AJ, Tillmann E, Subramanian S, Lehmkuhl L, Funkat AK, Leontyev S, Doenst T, Walther T, Gutberlet M, Mohr FW. Visceral arterial compromise during intra-aortic balloon counterpulsation therapy. Circulation. 2010 Sep 14;122(11 Suppl):S92-9. doi: 10.1161/CIRCULATIONAHA.109.929810. PMID 20837932
- [Background] Weber KT, Janicki JS. Intraaortic balloon counterpulsation. A review of physiological principles, clinical results, and device safety. Ann Thorac Surg. 1974 Jun;17(6):602-36. doi: 10.1016/s0003-4975(10)65706-2. No abstract available. PMID 4601521